CLINICAL TRIAL: NCT06771479
Title: A Randomized, Double-blind, Placebo-controlled Phase I Clinical Trial Evaluating the Safety and Immunogenicity of MVA Strain Monkeypox Attenuated Live Vaccine for Individuals Aged 18 and Above
Brief Title: A Study Evaluating the Safety and Immunogenicity of MVA Strain Monkeypox Attenuated Live Vaccine
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SIBP-V08-Ⅰ
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-01

CONDITIONS: Monkeypox
Keywords: Monkeypox vaccine; safety; vaccine; immunogenicity; Monkeypox
MeSH Terms: conditions — Mpox, Monkeypox

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Experimental group 1 (Experimental): Participants without a history of immunization against smallpox
  Interventions: Biological: MVA strain monkeypox attenuated live vaccine (low dose)
- Experimental group 2 (Experimental): Participants without a history of immunization against smallpox
  Interventions: Biological: MVA strain monkeypox attenuated live vaccine (high dose)
- Experimental group 3 (Experimental): Participants with a history of immunization against smallpox
  Interventions: Biological: MVA strain monkeypox attenuated live vaccine (low dose)
- Experimental group 4 (Experimental): Participants with a history of immunization against smallpox
  Interventions: Biological: MVA strain monkeypox attenuated live vaccine (high dose)
- Control group 1 (Placebo Comparator): Participants without a history of immunization against smallpox
  Interventions: Other: Placebo
- Control group 2 (Placebo Comparator): Participants with a history of immunization against smallpox
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: MVA strain monkeypox attenuated live vaccine (low dose) — Low dose MVA strain monkeypox attenuated live vaccine
  Arms: Experimental group 1; Experimental group 3
Biological: MVA strain monkeypox attenuated live vaccine (high dose) — High dose MVA strain monkeypox attenuated live vaccine
  Arms: Experimental group 2; Experimental group 4
Other: Placebo — Vaccine excipient
  Arms: Control group 1; Control group 2

SUMMARY:
This is a randomized, double blinded, controlled phase I clinical study. To evaluate the safety and immunogenicity of receiving two doses of MVA strain monkeypox attenuated live vaccine in individuals aged 18 years and above.

DETAILED DESCRIPTION:
This is a randomized, double blinded, controlled phase I clinical study. The study plans to recruit 120 participants aged 18 years and above. The experimental vaccine MVA strain monkeypox attenuated live vaccine has two different doses (low dose and high dose). The ratio of low-dose experimental group, high-dose experimental group, and placebo group is 1:1:1. Participants will be divided into three groups: healthy individuals, men who have sex with men, and HIV infected individuals, with a ratio of 2:1:1. Different groups will be divided into individuals with a history of vaccination against smallpox and those without a history of immunization, based on whether each population has a history of vaccination against smallpox. Each participant will receive one dose of the experimental vaccine or placebo on day 0 and day 28, respectively.

ELIGIBILITY:
Inclusion Criteria:

* On the day of enrollment, individuals aged 18 years or older with a history of smallpox vaccination must have been born before 1980;
* Can provide legal proof of identity;
* Be able to understand the experimental procedure and sign a written informed consent form, expressing agreement to participate in the experiment;
* Be able to participate in all planned follow-up visits and comply with all trial procedures (such as completing diary/contact cards and being able to return for visits);
* On the day of enrollment, the body temperature was less than 37.3 ℃ (axillary temperature);
* Men and women of childbearing age who have no plans to have children within 6 months and agree to take effective contraceptive measures within 6 months after receiving the experimental vaccine.

Exclusion Criteria:

* Individuals with a history of smallpox, monkeypox, or close contact with monkeypox in the past;
* Individuals who are allergic to any ingredients of eggs, vaccines, or substances used in production processes, or have a history of other severe allergies;
* Use immunoglobulin and/or any blood products within 3 months prior to administering the trial vaccine, or plan to use them during the trial period;
* Currently using salicylate drugs or planning long-term use during the trial period;
* Have used any experimental or unregistered products within one month prior to administering the trial vaccine, or plan to use them during the trial period;
* Administer inactivated vaccine within 14 days before administering the experimental vaccine or attenuated live vaccine within 30 days before administering the experimental vaccine;
* Chronic disease patients are in the acute or progressive phase of chronic disease;
* Long term use of immunosuppressants or other immunomodulatory drugs within 6 months prior to vaccination with the experimental vaccine;
* Having undergone chemotherapy or radiation therapy or organ and bone marrow transplantation related treatments for cancer or other diseases;
* Diseases or medical measures that lead to immune dysfunction, such as congenital immunodeficiency, organ and bone marrow transplantation, leukemia, lymphoma, Hodgkin's disease, multiple myeloma or malignant tumors, etc;
* Moderate or severe acute illness/infection, or febrile illness on the day of vaccination;
* Individuals with a history of thrombocytopenia or other coagulation disorders may be contraindicated for subcutaneous injection;
* Suffering from serious cardiovascular disease, serious liver and kidney disease, and diabetes that cannot be controlled by drugs;
* Previous history of mental or neurological disorders or family history;
* Currently suffering from various infectious, suppurative, and allergic skin diseases;
* Women of childbearing age: pregnant or lactating, or with a positive blood pregnancy test;
* Plan to move before the end of the trial or leave the local area for a long time during the scheduled trial visit;
* Abnormal blood routine, blood biochemistry, urine routine, electrocardiogram or heart disease related indicators before vaccination (except for minor abnormalities judged by doctors to have no clinical significance);
* Researchers believe that any situation that may affect the evaluation of the experiment;
* Active tuberculosis patients;
* For HIV infected individuals, the plasma HIV-1 RNA level during screening should be ≥ 200 copies/mL, or positive test for hepatitis B, hepatitis C and syphilis;
* For healthy people and men and women who have sex with each other, hepatitis B, hepatitis C, syphilis and HIV) are positive;
* Individuals who experience severe allergic reactions after the first dose of vaccination;
* Serious adverse events that are definitely related to the first dose of vaccination;
* For those who are newly discovered or occur after the first dose of vaccination and do not meet the inclusion criteria or the exclusion criteria for the first dose, the researcher shall determine whether to continue participating in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Immediate adverse events | 60 minutes after each dose of vaccination
  The occurrence of any adverse events within 60 minutes after each dose of vaccine immunization.
Solicited Adverse Events | 14 days after each dose of vaccination
  Adverse events defined by the protocol that occurred to the participant during 0-14 days after each dose of vaccination.
Unsolicited Adverse Events | 28 or 30 days after each dose of vaccination
  Other adverse events that occurred among participants within 0-28/30 days after each vaccination, in addition to the solicited adverse events.
Abnormal incidence rate of electrocardiogram | 14 days after each dose of vaccination
  Abnormal electrocardiogram after 14 days of vaccination with each dose.
Serious Adverse Events (SAE) | 12 months after the last dose
  That is serious adverse events, any serious adverse events that occurred to the participant during the study period.
Adverse Event of Special Interest (AESI) | 12 months after the last dose
  Adverse events that require special attention as specified in the experimental protocol.

OTHER OUTCOMES:
Geometric Mean Titer (GMT) of neutralizing antibodies | 14 days after the first dose of vaccine, before the second dose of vaccine and14 days, 28 days, 6 months, and 12 months after the second dose
  GMI of neutralizing antibodies against monkeypox virus in the experimental vaccine groups and the placebo group.
Seroconversion rate of neutralizing antibodies | 14 days after the first dose of vaccine, before the second dose of vaccine and14 days, 28 days, 6 months, and 12 months after the second dose
  The neutralizing antibody seroconversion rate against monkeypox virus in the experimental vaccine groups and the placebo group.
Seropositive rate of neutralizing antibodies | 14 days after the first dose of vaccine, before the second dose of vaccine and14 days, 28 days, 6 months, and 12 months after the second dose
  The neutralizing antibody seropositive rate against monkeypox virus in the experimental vaccine groups and the placebo group.
GMT of binding antibody | 14 days after the first dose of vaccine, before the second dose of vaccine and14 days, 28 days, 6 months, and 12 months after the second dose
  GMI of binding antibody against monkeypox virus in the experimental vaccine groups and the placebo group.
Seroconversion rate of binding antibody | 14 days after the first dose of vaccine, before the second dose of vaccine and14 days, 28 days, 6 months, and 12 months after the second dose
  The binding antibody seroconversion rate against monkeypox virus in the experimental vaccine groups and the placebo group.
Seropositive rate of binding antibody | 14 days after the first dose of vaccine, before the second dose of vaccine and14 days, 28 days, 6 months, and 12 months after the second dose
  The binding antibody seropositive rate against monkeypox virus in the experimental vaccine groups and the placebo group.
Cellular immune level | 14 days after the first dose of vaccine, before the second dose of vaccine and14 days, 28 days after the second dose
  Cellular immune levels of participants after receiving the experimental vaccine or placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Shuang Li, Master, Principal Investigator — Henan Infectious Disease Hospital; Qingxia zhao, Bachelor, Principal Investigator — Henan Infectious Disease Hospital
Locations (1):
- Henan Infectious Disease Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No